CLINICAL TRIAL: NCT03711968
Title: Interoception and Sense of Movement in the Patient With Multiple Sclerosis: Proposal of a Rehabilitation Protocol
Brief Title: Interoception and Sense of Movement in the Patient With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, Medical Doctor, University of Roma La Sapienza
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 5125
Record Dates: First submitted 2018-10-14; First posted 2018-10-19 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: Interoception; Sense of movement; Posture; body scheme
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): Rehabilitative treatment protocol:
  Therapeutic exercise 8 mono-weekly sessions, 5 patients per group, duration 60 minutes and two sessions of single treatment, duration 60 minutes (duration of treatment about two months, considering also any recovery sessions)
  Interventions: Other: Rehabilitative treatment protocol
- Waiting list (No Intervention): Intervention: The WL patients will be taken into the same treatment at the end of the experimental protocol, after T2 evaluation. In this period they act like a control group.

INTERVENTIONS:
Other: Rehabilitative treatment protocol — A combination of: postural exercise with visual spatial tasks, relaxation, balance exercise, motricity improvement and cognitive rehabilitation.
  Arms: Treatment group

SUMMARY:
To evaluate the effectiveness of an experimental rehabilitative protocol with specific tasks for the improvement of body awareness and the motor scheme in the patient with multiple sclerosis (EDSS <2.5).

Primary outcome: improvement of the interoception (awareness of the body) and of the related motor capacity Secondary outcomes: improvement of balance and postural self-correction control

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronically progressive, disabling, autoimmune disease that affects the central nervous system causing a wide spectrum of sensory, motor, and neuropsychiatric signs and symptoms. In the great part of patients with MS, there is a cognitive deficit that can start already in the early stages of the disease. Disability related to the disease is usually investigated through the Expanded Disability Status Scale (EDSS), however, the scale does not evaluate some very disabling aspects of the disease such as diplopia, fatigue and the impact of cognitive disorders.

The posture and postural self-correction are dependent on the image that anyone have of his own body and on the perception of it in the space, both internal and external. In multiple sclerosis proprioception and interoception are often altered due to motor and cognitive impairment.

The investigators propose a rehabilitative protocol that combine postural rehabilitation with specific visual-spatial tasks, relaxation sessions with self-awareness improvement and cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* BMI<30
* Diagnosis of multiple sclerosis for less than 10 years
* Course of relapsing remitting type
* Relapse-free for at least 30 days
* EDSS score <2,5
* FDA-approved disease-modifying therapy for at least 6 months
* MMSE>24
* Public health guidelines for participating in physical activity

Exclusion Criteria:

* Other concurrent neurological and psychiatric diseases (like schizophrenia, bipolar disorder I or II and substance abuse disorders)
* Oncological diseases
* Cardiovascular disease, pacemaker carrier
* Diabetes
* Rheumatological diseases
* Scoliosis >20° Cobb
* Previous surgery on the spine
* Pregnancy
* Other physiotherapy in progress

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Change in interoception | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  Multidimensional Assessment of Interoceptive Awareness (MAIA) total score minimum 0 - 40 obtained by sum of the 8 subscales: noticing 0 - 5, not distracting 0 - 5, not worring 0 - 5, attention regulation 0 - 5, emotional awareness 0 - 5, self regolation 0 - 5, body listening 0 - 5, Trusting 0 - 5. Higher values represent a better outcome.

SECONDARY OUTCOMES:
Change in posture | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  Clinical assessment of spinal curve in normal posture and in self correction of posture.
Change in balance 1 | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  Tinetti balance assessment tool. Total score 0 - 28 obtained by sum of 2 section: balance section 0 - 16, Gait section 0 - 16. Higher values represent a better outcome.
Change in balance 2 | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  Baropodometry in normal posture and in self correction of posture.
Change in QOL. | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  The Short Form (12) Health Survey. The 12 questions includes one of two items from each of eight health concepts: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE) and Mental Health (MH). Two synthetic indices are obtained by a special software, Physical component summary (PCS - 12) score 18.4 - 57.8 and Mental component summary (MCS - 12). score 18.7 - 65.2. Higher values represent a better outcome.
Change in body image 1 | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  Body Image Scale (BIS). Total score 0 - 30 obtained by the sum of 10 items 0 - 3, lower values represent a better outcome.
Change in body image 2 | At the end of the cycle 1 (60 days), and at follow-up (120 days)
  Trunk Appearance Perception Scale (TAPS). The TAPS includes 3 sets of figures that depict the trunk from 3 viewpoints: looking toward the back, looking toward the head with the patient bending over, and looking toward the front. This last view has two sets of drawings, one for males and one for females. Each drawing is scored from 1 (greatest deformity) to 5 (smallest deformity) and a mean score is obtained by adding the scores for the 3 drawings and dividing by 3. Higher values represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Valter Santilli, MD, Study Director — University of Roma La Sapienza
Locations (1):
- Umberto I Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided